CLINICAL TRIAL: NCT06662370
Title: Remplacement de l'œsophage Par Une Greffe d'œsophage Humain décellularisé
Brief Title: Esophageal Replacement With a Decellularized Human Esophagus Graft
Acronym: ESOGRAFT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP220793
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Stenosis
Keywords: Tissue engineering; Esophageal replacement; Esophageal stenosis; Caustic injury; Radiotherapy; Anastomotic stenosis; Esophageal stent
MeSH Terms: conditions — Esophageal Stenosis

STUDY DESIGN:
Intervention Model Description: Open-label, non-comparative, phase I/II, single-arm, multicenter trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Esophagus replacement (Experimental)
  Interventions: Other: Replacement of the esophagus with a decellularized human esophagus graft

INTERVENTIONS:
Other: Replacement of the esophagus with a decellularized human esophagus graft — The Decellularized Human Esophagus (DHE) will be surgically implanted under general anesthesia via right or left thoracotomy or cervicotomy, depending on the location of the stenosis, to replace the esophageal defect created by resection of the stenosis. An omentoplasty is performed laparoscopically beforehand to provide secondary coverage of the graft area. A temporary esophageal stent is placed endoscopically to cover the DHE and the two anastomoses for a period of 3 months, to prevent the development of an anastomotic fistula and stenosis of the graft area.

SUMMARY:
The aim of the study is to analyze over a 12 month-period, the safety and the efficacy of a circumferentiel oesophageal replacement of the esophagus by a decelularized human esophagus, in 24 patient with a short esophageal stenosis refractory to endoscopic dilatations.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65
* Caustic, traumatic, anastomotic, post-operative, radiation-induced or post-endoscopic (mucosal resection, submucosal dissection) benign esophageal stricture refractory to endoscopic dilatation.
* For women: effective contraception for the entire duration of the study (from signature of consent to end of follow-up)
* Affiliated or beneficiary of a social security scheme.
* Free written consent signed by the participant and the investigator.

Exclusion Criteria:

* Weight loss > 10% of body weight over last 3 months
* Stenosis > 5 cm in length
* Multiple strictures
* Esophageal mouth stenosis
* Anterior surgery close to the operative zone
* Complete anterior omentectomy
* Tumour stenosis or progressive tumour pathology
* Non-stabilized psychiatric disorders
* Participation in another interventional study
* Pregnant or breast-feeding women
* Women of childbearing age without effective contraceptive measures:

All women of childbearing age must have a negative pregnancy test prior to treatment and must agree to maintain highly effective contraception using contraceptive measures from the date of consent until 12 months due to the risks associated with anesthesia during endoscopy

* Uncontrolled sepsis
* Related to the transplant procedure

  * ASA score ≥ 3,
  * Severe respiratory insufficiency (FEV1 < 1 L),
  * Decompensated hepatic cirrhosis or presence of esophageal varices,
  * Chronic renal insufficiency (creatinine > 1.25 N),
  * Myocardial infarction less than 6 months old or progressive heart disease,
  * WHO general condition > 2,
  * Weight loss >20% not recovered after renutrition.
* Contraindication to general anaesthesia, analgesics and antibiotics.
* Conditions requiring long-term immunosuppressive or corticosteroid treatment.
* Patients under curatorship or guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Morbidity/mortality | At 3 months after surgery
  Safety criterion : morbidity/mortality defined by :
  Refractory stenosis, leaking, sepsis, stent migration, death, complete rupture of anastomoses, uncontrolled mediastinal sepsis requiring removal of the substitute and/or esophagectomy, delamination of the tissue graft, tracheobronchial wound intra-operatively or oesotracheal fistula postoperatively, upper digestive obstruction after stent removal preventing any attempt to dilate the graft zone, or upper digestive obstruction after stent removal preventing any attempt to dilate the graft zone
Nutritional autonomy | At 12 months after esophageal replacement
  Efficacy criterion: nutritional autonomy at 12 months after esophageal replacement defined as stable weight with exclusive oral nutrition and without esophageal stenting for at least 3 months, and without persistent symptomatic scar stenosis after 5 endoscopic dilatation sessions

SECONDARY OUTCOMES:
Safety of the procedure | At 12 months after esophageal replacement
  The morbidity and mortality of the procedure will be defined by the occurrence of a complication such as leakage, sepsis, recurrent paralysis, esophageal stricture refractory to dilatation, anastomotic fistula, sepsis, esophageal perforation, cardio-respiratory complication (pneumopathy, pleural effusion, pulmonary embolism, AC/FA, infarction), death, tissue graft disintegration, postoperative tracheobronchial wound or oesotracheal fistula, or upper digestive obstruction after stent removal preventing any attempt to dilate the graft zone), for 12 months from the date of surgery.
Presence of complete re-epithelialization, and integration into the native esophagus | At 3 months after surgery
  Assessed by endoscopy
Presence of complete re-epithelialization, and integration into the native esophagus | At 12 months after surgery
  Assessed by CT scan with gel ingestion and intravenous contrast injection
Normal bolus transit | At 6 months after surgery
  Assessed by barium deglutition
Normal bolus transit | At 12 months after surgery
  Assessed by barium deglutition
Esophageal manometry | At 12 months after surgery
Percentage of procedures interrupted for logistical reasons | Up to 14 months
  Logistical reasons are defined as :
  * An incident during transport from the Human Tissue Bank to the operating room, resulting in the loss of the graft
  * Accidental rupture of graft packaging, with risk of loss of sterility
  * An incident occurring during the graft thawing procedure
Overall survival and Safety of procedure | At 12 months after surgery
  Patient survival at 12 months regardless of cause of death
Impact of procedure on quality of life | At 6 months after surgery
  EORTC QLQ-OG25 module Score varying between 25 and 100, the higher the score the more severe the symptoms
Impact of procedure on quality of life | At 12 months after surgery
  EORTC QLQ-OG25 module Score varying between 25 and 100, the higher the score the more severe the symptoms
Impact of procedure on quality of life | At 6 months after surgery
  SF12V2 modules It is a 12 items score varying from to 0 to 100. The higher the score, the better the quality of life
Impact of procedure on quality of life | At 12 months after surgery
  SF12V2 modules It is a 12 items score varying from to 0 to 100. The higher the score, the better the quality of life
Estimating the cost of the procedure for one patient | At 12 months
  -Direct medical costs of the procedure: constitution (tissue engineering), storage and transport of the esophageal stent, hospital stay for graft surgery, emergency room visits, scheduled or unscheduled re-hospitalizations, follow-up in hospital consultations, scheduled or unscheduled outpatient physician visits, outpatient biological procedures, outpatient medical imaging, drug prescriptions, transport and coordination time by the expert team.
Estimating the cost of the procedure for target population | At 12 months
  -Simulation using trial data of costs for all patients with esophageal transplant indication

IPD SHARING:
Plan to Share IPD: Undecided